CLINICAL TRIAL: NCT02804009
Title: Evaluating and Predicting Anxiety in Patients Undergoing Elective Coronary Angiography
Brief Title: Elective Coronary Angiography and Anxiety Study
Acronym: ANGST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: General and Teaching Hospital Celje (Other)
Collaborators: University Psychiatric Clinic Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: GenealTHC
Record Dates: First submitted 2016-06-09; First posted 2016-06-17 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-06

CONDITIONS: Anxiety
Keywords: anxiety; coronary angiography
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Anxiety will be assessed from two aspects, the somatic and emotional. ANGST aims to determine how anxiety correlates with psychological parameters (personality traits, coping strategies and depressive symptoms) and with the outcome of elective coronary angiography (CA).

DETAILED DESCRIPTION:
This research is a prospective cross-section study of patients undergoing elective CA. Research design will allow studying anxiety at four timepoints and its correlation with CA outcome and psychological parameters. This study will be conducted at the Coronary care unit of the department of Cardiology, General and Teaching Hospital Celje, Slovenia.

Data regarding prior to CA, during hospital stay and after discharge variables will be collected in order to control for confounding variables when testing the association between anxiety and psychological parameters. All the data needed for this study will be collected within one month from the patient enrollment in this study at four occasions: (1) 14 days prior CA - all patients will receive questionnaires by post, (2) on the day of the admission, 2-4 hours before CA, (3) 24 hours after CA, but prior to discharge and (4) 4-6 weeks after discharge. Clinical and demographical data will be collected from medical records. Data regarding anxiety and other psychological parameters will be assessed using standardized questionnaires. These will be sent to the patient together with covering letter providing instructions to complete the questionnaires 14 days prior CA without help of family members/friends. A month after CA, the questionnaires for anxiety and depressive symptoms will be sent to participants address with reply paid envelope provided.

The Republic of Slovenia National Medical Ethics Committee has approved this study.

ELIGIBILITY:
Inclusion Criteria:

* invited to elective CA because of suspected/unknown: coronary artery disease, valvular heart disease, heart failure etiology, unexplained arrhythmia, cardiomyopathy etiology;
* written consent;
* completed first set of questionnaires 14 days prior to coronary angiography

Exclusion Criteria:

* need for an urgent coronary angiography,
* coronary angiography in last 6 months,
* unable to provide written consent,
* severe physical and/or mental disease/disability,
* help needed in completing the questionnaires,
* unsigned consent form,
* incomplete first set of questionnaires 14 days prior to coronary angiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are invited to elective coronary angiography due to suspected/unknown: coronary artery disease, valvular heart disease, heart failure etiology, unexplained arrhythmia, and cardiomyopathy etiology.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change between emotional anxiety in patients without depressive symptoms | Baseline, 2 hours before CA, 24h after CA and 1 month after CA
  Measured with Spielberger State Anxiety Inventory
Change between somatic anxiety in patients without depressive symptoms | Baseline, 2 hours before CA, 24h after CA and 1 month after CA
  Measured with Beck Anxiety Inventory

SECONDARY OUTCOMES:
Depressive symptoms | Baseline, 1 month after CA
  Measured with Cardiac Depression Scale
Personality traits | Baseline
  Measured with 10-item short version of Big Five Inventory
Response on stress | Baseline
  Measured with COPE Inventory
Trait Anxiety | Baseline
  Measured with Spielberger Trait Anxiety Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Mitja Lainščak, MD, PhD, Study Director — Professor of Internal Medicine, General and Teaching Hospital Celje
Locations (1):
- General and Teaching Hospital Celje, Celje, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trotter R, Gallagher R, Donoghue J. Anxiety in patients undergoing percutaneous coronary interventions. Heart Lung. 2011 May-Jun;40(3):185-92. doi: 10.1016/j.hrtlng.2010.05.054. Epub 2010 Aug 17. PMID 20723986
- [Background] Astin F, Jones K, Thompson DR. Prevalence and patterns of anxiety and depression in patients undergoing elective percutaneous transluminal coronary angioplasty. Heart Lung. 2005 Nov-Dec;34(6):393-401. doi: 10.1016/j.hrtlng.2005.05.002. PMID 16324958
- [Background] Tully PJ, Cosh SM, Baumeister H. The anxious heart in whose mind? A systematic review and meta-regression of factors associated with anxiety disorder diagnosis, treatment and morbidity risk in coronary heart disease. J Psychosom Res. 2014 Dec;77(6):439-48. doi: 10.1016/j.jpsychores.2014.10.001. Epub 2014 Oct 14. PMID 25455809
- [Background] Pedersen SS, Denollet J, Spindler H, Ong AT, Serruys PW, Erdman RA, van Domburg RT. Anxiety enhances the detrimental effect of depressive symptoms on health status following percutaneous coronary intervention. J Psychosom Res. 2006 Dec;61(6):783-9. doi: 10.1016/j.jpsychores.2006.06.009. PMID 17141666
- [Background] Vogelzangs N, Seldenrijk A, Beekman AT, van Hout HP, de Jonge P, Penninx BW. Cardiovascular disease in persons with depressive and anxiety disorders. J Affect Disord. 2010 Sep;125(1-3):241-8. doi: 10.1016/j.jad.2010.02.112. Epub 2010 Mar 12. PMID 20223521
- [Background] Damen NL, Versteeg H, Boersma E, de Jaegere PP, van Geuns RJ, van Domburg RT, Pedersen SS. Indication for percutaneous coronary intervention is not associated with symptoms of anxiety and depression. Int J Cardiol. 2013 Oct 12;168(5):4897-8. doi: 10.1016/j.ijcard.2013.07.022. Epub 2013 Jul 19. No abstract available. PMID 23871630
- [Background] van Gestel YR, Pedersen SS, van de Sande M, de Jaegere PP, Serruys PW, Erdman RA, van Domburg RT. Type-D personality and depressive symptoms predict anxiety 12 months post-percutaneous coronary intervention. J Affect Disord. 2007 Nov;103(1-3):197-203. doi: 10.1016/j.jad.2007.01.030. Epub 2007 Mar 7. PMID 17346801
- [Background] Chaudhury S, Srivastava K. Relation of depression, anxiety, and quality of life with outcome after percutaneous transluminal coronary angioplasty. ScientificWorldJournal. 2013 Nov 10;2013:465979. doi: 10.1155/2013/465979. eCollection 2013. PMID 24319368
- [Background] van den Berge JC, Utens EM, Dulfer K, Hartman EM, van Geuns RJ, Daemen J, van Domburg RT. Can anxiety and depression, separately or in combination predict subjective health status 10 years post-PCI? Int J Cardiol. 2015;186:57-9. doi: 10.1016/j.ijcard.2015.03.147. Epub 2015 Mar 17. No abstract available. PMID 25814344
- [Derived] Palandacic AK, Ucman S, Kovacic D, Sarotar BN, Lainscak M. Anxiety in patients referred for elective coronary angiography: a prospective cohort study. BMC Cardiovasc Disord. 2025 Dec 29. doi: 10.1186/s12872-025-05454-5. Online ahead of print. PMID 41457207